CLINICAL TRIAL: NCT01483235
Title: Design, Implementation and Evaluation of a Reduced Cardiac Rehabilitation Program
Brief Title: Reduced Cardiac Rehabilitation Program
Acronym: rCRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Simon Fraser University (Other)
Responsible Party: Principal Investigator, Alejandra Farias-Godoy, MD, MSc, PhD candidate. Principal Investigator, Simon Fraser University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 37553; 37553 (Other: Simon Fraser University)
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Cardiovascular Disease; Obesity; Dyslipidemia
Keywords: cardiac rehabilitation; prevention; exercise capacity
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reduced cardiac rehabilitation (rCRP) (Experimental): The rCRP is the intervention group, compared to the standard cardiac rehabilitation program group (sCRP). The rCRP will have the core elements of the sCRP, that is, in-hospital exercise sessions, dietary counseling, educational sessions, follow-up with the cardiologist, dietician and exercise specialist. The only difference will be the number of in-hospital exercise sessions (10 sessions for the rCRP v/s 32 sessions for the sCRP). Patients from rCRP will receive individual exercise guidelines, an educational package with questions of the week and a diary to record their exercise sessions (logbook), that will serve as a self-monitoring system.
  Interventions: Behavioral: Reduced cardiac rehabilitation group intervention (rCRP).
- Standard cardiac rehabilitation (sCRP) (Active Comparator): The standard cardiac rehabilitation (sCRP) follows the standard cardiac rehabilitation program model of a four-month period. Patients receive an initial intake evaluation by a cardiologist, nurse, exercise specialist and dietitian before starting the program. The program consists of 32, twice weekly in-hospital exercise sessions, educational sessions, nutritional counseling, medical care, psychological screening and smoking cessation if needed.
  Interventions: Behavioral: Standard cardiac rehabilitation intervention

INTERVENTIONS:
Behavioral: Reduced cardiac rehabilitation group intervention (rCRP). — The rCRP is a comprehensive intervention that will keep the same nature of therapies as the standard cardiac rehabilitation group (sCRP). The difference with the sCRP resides in the number of hospital based exercise sessions; instead of 32 sessions there will be 10 sessions spread throughout the 4 months of intervention (hence, not a shorter program). The rCRP intervention works within the sCRP. Hence, those randomized to the rCRP will be supervised in the same facility and by the same clinical staff as those in the sCRP. Patients from rCRP will receive individual exercise guidelines, an educational package with questions of the week and a diary to record their exercise sessions (logbook), that will serve as a self-monitoring system.
  Other Names: rCRP
  Arms: Reduced cardiac rehabilitation (rCRP)
Behavioral: Standard cardiac rehabilitation intervention — The standard cardiac rehabilitation is a multidisciplinary four-month intervention to modify ischemic heart disease risk factors and lifestyle behaviours. These programs aim to reduce morbidity and mortality by improving adherence to regular physical activity, a healthy diet and smoking cessation, as well as risk factor modification. Patients receive an initial intake evaluation by a cardiologist, nurse,exercise specialist and dietitian before starting the program. The program consists of 32, twice weekly in-hospital exercise sessions, educational sessions, nutritional counselling, medical care, psychological screening and smoking cessation if needed.
  Other Names: sCRP
  Arms: Standard cardiac rehabilitation (sCRP)

SUMMARY:
Standard cardiac rehabilitation programs (sCRP) aim to improve risk factors for heart disease such as high blood pressure, weight control, exercise and diet in order to decrease the chances of having heart problems in the future. These programs decrease morbidity and mortality but face important challenges: 1) Long waiting lists to participate in these programs. For example, St. Paul's Hospital has an intake capacity of 480 patients per year. Patients usually wait one to three months to start the program. 2) There is a vast heterogeneity of patients within the same program, from those that have never experienced heart problems to those that have already had a heart attack, chest pain or stroke. Therefore, patients with different medical problems receive the same treatment. 3) Facilities can be inconveniently located which leads to transportation difficulties, 4) The program is time consuming and classes are held in working times, 5) Shortly after completion, patients seem to lose what they have gained in the program. These caveats need to be addressed to improve the efficacy, delivery and capacity of sCRP for the increasing population of patients with heart disease.

The investigators want to compare a reduced cardiac rehabilitation program (rCRP) with the standard cardiac rehabilitation program (sCRP) in patients with risk factors for heart disease as well as patients that already suffer from this condition, including those at higher risk. The rCRP will offer the same services as the sCRP; the only difference is the number of hospital based exercise sessions. While the sCRP offers 32 hospital based supervised exercise sessions, the rCRP will offer 10 hospital based exercise sessions. The rCRP would be a 'middle of the road alternative program' that would have the benefits of a hospital based program and the flexibility of a home based intervention. The rCRP would offer an alternative for patients that do not need constant supervision and would allow the sCRP health care team to focus on those patients who have more serious heart conditions. The rCRP would be a unique intervention because it integrates a less intensive cardiac rehabilitation into the pre-existing sCRP model. This alternative would help overcome the caveats of standard cardiac rehabilitation programs.

DETAILED DESCRIPTION:
This study is a two group randomized controlled trial, non-inferiority design, where the rCRP (intervention group) will be compared with the sCRP (control group). Eligible patients will be asked to participate in the study at the cardiac rehabilitation program intake clinic. Consenting participants will be asked to sign an informed consent and undergo a baseline assessment. This assessment will consist of a medical history, exercise capacity (stress test), blood test, blood pressure, anthropometric measurements, lifestyle behaviours and psychosocial measurements. The baseline assessment will be done before participants start the program. Consecutively, randomization will take place stratified according to gender to either the sCRP or rCRP. The same assessment called exit assessment will be performed at four to six months from baseline, at the cardiac rehabilitation program exit clinic (at program completion) and at 16 to 20 months from baseline (one year follow-up from cardiac rehabilitation program completion) to assess the immediate and sustainable effect, respectively.

The following research questions will be addressed:

1. Is the reduced cardiac rehabilitation program (intervention group) as effective as the standard cardiac rehabilitation program (control group) for improving exercise capacity and ischemic heart disease risk factors at both program completion (four to six months from baseline) and at one year from program completion (16 to 20 months from baseline)?
2. Will the reduced cardiac rehabilitation program have better adherence than the standard cardiac rehabilitation program?

ELIGIBILITY:
Inclusion Criteria:

1. Men and women (equal distribution) with risk factors for ischemic heart disease (primary prevention) or documented ischemic heart disease (secondary prevention) accepted in the cardiac rehabilitation program of St. Paul's Hospital.
2. Patients with documented ischemic heart disease (secondary prevention) classified as low and moderate risk according to the AACVPR risk stratification criteria for cardiac patients.

Exclusion Criteria:

1. Patients with documented ischemic heart disease (secondary prevention)at high risk according to the AACVPR risk stratification criteria for cardiac patients.
2. Patients will also be excluded if they have the following:

   * Uncontrolled metabolic factors (renal failure, uncontrolled diabetes, endocrinopathies
   * Scheduled revascularization
   * Unable to provide informed consent
   * Unlikely to survive due to non cardiac issues
   * Psychiatric conditions that would interfere with compliance.
   * Center for Epidemiologic Studies Depression scale higher than 16 points.
   * Those coming to the cardiac rehabilitation program due to congenital heart disease with no risk factors for ischemic heart disease.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2006-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | Data collection to be completed in September 2011
  Exercise capacity will be determined through a symptom-limited maximal treadmill exercise test using the Bruce protocol and reported as total time in seconds in the treadmill. Participants will undergo continuous 12-lead ECG monitoring during the test. Participants will have their baseline, exit(program completion) and one-year (16 to 20 months from baseline) exercise stress tests conducted at the ECG stress laboratory at St. Paul's Hospital.

SECONDARY OUTCOMES:
Metabolic risk factors. | Data collection to be completed by September 2011
  Total cholesterol, HDL-C, triglycerides and blood glucose will be assessed from fasting blood samples. The Friedewald equation will be used to calculate LDL-C. To assess for change in global risk score, the Framingham risk score and the Progression of Disease risk score will be used for primary and secondary prevention patients respectively. Blood pressure will be measured with a manual sphyngomanometer. These outcomes will be assessed at baseline (program intake), program completion (four to six months from baseline) and at 16 to 20 months from baseline.
Lifestyle | Data collection to be completed in September 2011
  Leisure time physical activity will be determined by the four-week modified Minnesota LTPA questionnaire and reported as the average weekly kilocalories (kcal/wk) expended through physical activity and exercise. Diet will be reported as percent daily kilocalories for fat, protein and carbohydrates using a three-day food record. Smoking status will be assessed by self-report. These outcomes will be measured at baseline (program intake), program completion (four to six months from baseline) and at 16 to 20 months from baseline.
Psychosocial measures | Data to be collected by September 2011
  Health related Quality of life will be assessed by the Euro Quality of Life questionnaire. Self-efficacy will be assessed with the self-efficacy questionnaire that has two components: a general self-efficacy assessment and exercise-specific assessment. These outcomes will be measured at baseline (program intake), program completion (four to six months from baseline)and at 16 to 20 months from baseline.
Anthropometry | Data to be collected by September 2011
  Body mass index will be calculated from weight in kilograms divided by height in metres squared. Waist circumference will be recorded in centimetres, taken at the point of maximal narrowing following a normal expiration. Hip circumference will be recorded in centimetres taken at the point of maximal gluteal protuberance. Waist to hip ratio will be calculated by simple division. These outcomes will be measured at baseline (program intake), program completion (four to six months from baseline) and at 16 to 20 months from baseline.
Program adherence | Data collection to be completed in September 2011
  Assessed as percent attendance to in-hospital sessions. Overall physical activity adherence will be assessed with the LTPA questionnaire measured as weekly kilocalorie/week expended. This outcome will be measured at baseline (program intake), at program completion (four to six months from baseline)and at 16 to 20 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Lear, PhD, Principal Investigator — Simon Fraser University; Alejandra Farias-Godoy, MD, MSc, Principal Investigator — Simon Fraser University
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada